CLINICAL TRIAL: NCT06731127
Title: Vaccines in a Time of Dual Pandemic: COVID-19 Vaccine in People With HIV
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Mario Ostrowski, Clinical Professor, University of Toronto
Other Study IDs: 40713
Record Dates: First submitted 2024-12-03; First posted 2024-12-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- People with HIV (PWH) Immune responders (n=35): undetectable viral load for 1+ year, CD4 >500/uL, CD4/CD8 ratio >1 including individuals with a historical, low CD4 nadir
- People with HIV (PWH) Immune non-responders (n= 10): undetectable viral load, CD4 <350/uL or CD4/CD8 ratio <0.75 for 1+ year
- People with HIV (PWH) Low-level viremics (n= 10): low-level viremia (<1,000 copies/mL) for 1+ year, any CD4, any CD4/CD8 ratio
- HIV-negative control (n= 20): age and sex matched

SUMMARY:
This is a prospective, non-randomized observational study to examine SARS-CoV-2 vaccine immunogenicity, immune activation and HIV reservoirs in people with HIV infection in comparison with HIV-negative individuals, in those aged 55 or more.

As Canada is currently rolling out COVID-19 vaccines, the two most imminent vaccines are mRNA vaccines. These are the Pfizer-BioNTech COVID-19 vaccine given 3 weeks apart and the Moderna COVID-19 vaccine given 4 weeks apart. Given the unique storage requirements of these vaccines, it is expected that the Moderna vaccine will be used primarily in primary care clinics such as Maple Leaf Medical Clinic, Toronto. However, the protocol will also allow observational study of individuals being administered with the Pfizer-BioNTech vaccine if it is also available. The investigators predict general availability of both vaccines to the primary care population by March 1, 2021. Vaccination will occur as per clinical and public health guidelines. COVID-19 vaccines will not be administered as a part of this research study. This is a single site longitudinal study where 75 participants in total are followed over 48 weeks with blood draws and saliva sampling. The breakdown of study arms is described here:

• PWH Immune responders (n= 35): undetectable viral load for 1+ year, CD4 >500/uL, CD4/CD8 ratio >1 including individuals with a historical, low CD4 nadir

• PWH Immune non-responders (n= 10): undetectable viral load, CD4 <350/uL or CD4/CD8 ratio <0.75 for 1+ year

• PWH Low-level viremics (n= 10): low-level viremia (<1,000 copies/mL) for 1+ year, any CD4, any CD4/CD8 ratio

• HIV-negative control (n= 20): age and sex matched

DETAILED DESCRIPTION:
People with HIV (PWH) may experience an increased risk of COVID-19 related diseases or mortality upon SARS-CoV-2 infection1-5, and COVID-19 vaccines will play a significant role in combating the pandemic. Currently, there are two mRNA vaccines to be utilized in Ontario (Pfizer-BioNTech, Moderna), both with a two-dose regimen6,7. While data so far do not suggest any particular safety concerns for PWH, only a limited number of PWH have participated in COVID-19 vaccine trials, and they were recruited late during two recent large confirmatory approval studies. In addition, emergency approval review of the confirmatory trials for one of the vaccines did not include PWH in safety and efficacy calculations7,8, including PWH receiving antiretroviral therapy (ART) who present ongoing low-level viremia, immunosenescence and/or persistent immune activation. Nevertheless, PWH are encouraged to get vaccinated promptly while data collection continues.

A significant gap in our knowledge - and based on experience with vaccines administered to PWH for other pathogens9 - is whether COVID-19 vaccines may have any impact on ongoing chronic inflammation and other immune dysregulation that can exacerbate co-morbidity incidence or affect the dynamics of the human immunodeficiency virus (HIV) reservoir. Therefore, understanding how COVID-19 vaccines affect immune activation and HIV reservoirs in PWH is of paramount importance and may have implications for 38 million PWH globally. Furthermore, premature immunosenescence previously reported in PWH coupled with the heterogeneity of immune reconstitution following initiation of ART suggests that it will be crucial to determine whether COVID-19 vaccines can induce protective and robust immune responses both in the short-term and long-term, particularly in specific subgroups with diminished immunocompetence. Elucidating the effect of COVID-19 vaccines on immune activation and HIV reservoir as well as vaccine efficacy in PWH are critical but are unlikely to be evaluated by vaccine sponsors.

The investigators expect that our study population will not be included in the early priority administration of the COVID-19 vaccines in Ontario. Our target population is PWH over 55 of age often with comorbidities, who are likely to be offered vaccination within a most opportune window and convenient timeframe for this directed research.

Risk of COVID-19 in people with HIV (PWH)

Although data on the risk of COVID-19 on people with HIV (PWH) are limited, emerging evidence suggests that PWH may experience an increased risk of COVID-19 related diseases or mortality upon SARS-CoV-2 infection. For instance, a prospective observational study from the United Kingdom showed that after adjusting for several variables including sex, ethnicity, age and selected comorbidities, HIV-positive status remained significantly associated with an increased risk of day-28 mortality among individuals hospitalized for COVID-195. Another study from the United Kingdom also showed that PWH experience enhanced risk of COVID-19 mortality after adjusting for age, sex, deprivation, ethnicity, smoking and obesity (adjusted hazard ratio 2.59; 95% CI 1.74-3.84)3. Likewise, a population cohort study from South Africa also demonstrated that HIV is associated with COVID-19 mortality with an adjusted hazard ratio of 2.14 (95% CI 1.70-2.70)10. It is important to note, however, that several potential confounders were not included in these studies such as occupation and surrogate markers of HIV control11.

Meanwhile, other studies suggest a more nuanced role HIV may play in COVID-19 outcomes. For example, while a study from New York showed that a higher proportion of PWH experienced hospitalization, intensive care unit (ICU) admission and/or death due to COVID-19 as compared to HIV-negative individuals, the authors commented that most PWH who experienced poor COVID-19 related outcomes had lower (< 500 cells/uL) CD4 count12. Similarly, a multinational study found that a lower (< 200 cells/mm3) CD4 count is associated with severe outcomes as defined by ICU admission, mechanical ventilation or death13. Another multicenter cohort study involving three European countries conducted a multivariate analysis to show that the only factor associated with severe COVID-19 is a current CD4 count of less than 350 cells/uL (aOR 2.85; 95% CI 1.26-6.44), and with mortality, a low nadir CD4 T cell count4. In sum, immunodeficiency may be a possible risk factor for COVID-19 disease severity in PWH in the context of viral suppression. Vaccine-mediated prevention of SARS-CoV-2 infection and/or severe disease with COVID-19 is essential in this vulnerable population.

COVID-19 vaccines will play a significant role in combating the pandemic. Currently, there are two mRNA vaccines to be utilized in Ontario (Pfizer-BioNTech, Moderna), both with a two-dose regimen.

Current National Advisory Committee on Immunization (NACI) recommendation states that "no safety signals of concern have been noted to date in non-immunosuppressed participants with an immunocompromising condition (e.g., stable HIV infection) included in the clinical trials" and that "people living with HIV that are considered immunocompetent may be vaccinated"15. However, the number of PWH recruited in these trials to date is very small. There is also some suggestion that older age and its associated immunosenescence may have important implications as evidenced by the trial results of reduced vaccine efficacy with a wide confidence interval in older (aged 65+) participants. To the extent older PWH are often characterized as susceptible to accelerated or accentuated signs of aging and immunosenescence, those findings underline the need to evaluate vaccine effects more clearly in this group. Otherwise, vaccine efficacy in particular PWH subsets including those with ongoing low-level viremia, immunosenescence and/or persistent immune activation is largely unknown.

Immunogenicity At this time, vaccines that can elicit robust and long-lasting responses from T cells and B cells are presumed to be immune correlates of protection in vaccinated individuals16. Both the Pfizer-BioNTech and Moderna vaccines have described immunogenicity in their earlier trials.

Data on immunogenicity and potential correlates of protection are limited at this time and lacking in PWH, especially in subsets with suboptimal immune restoration. Given the gaps in vaccine approval analysis for PWH, it is important to establish immunogenicity profiles in PWH receiving vaccines.

Persistent immune activation in PWH

Despite the incredible advances in the effectiveness of ART, viral suppression with ART is often insufficient to completely dampen the heightened immune activation present in PWH. Importantly, persistent immune activation and/or inflammation have emerged as independent predictors of morbidity and mortality in ART-treated PWH. Key markers of immune activation and inflammation in the context of HIV infection include plasma levels of IL-6 and C-reactive protein (CRP) as well as the coagulation marker D-dimer and soluble monocyte activation marker sCD1420-22. Another widely used marker of inflammation is T cell activation as defined by the expression of CD38 and HLA-DR23.

Immune activation evidently has a negative impact on the morbidity and mortality of PWH, but it has also been linked to the HIV reservoir24. The implications of the COVID-19 vaccines on immune activation, and in turn, on the HIV reservoir of ART-treated PWH remain unclear. Given the lack of evidence in COVID-19 vaccines, our current understanding of their potential impact on PWH can only be extrapolated from previous studies on non-COVID-19 vaccines.

Non-COVID-19 vaccines and their effect on PWH

There are several non-COVID-19 vaccines which are recommended for adult PWH in Canada, including those against influenza, tetanus/diphtheria/whooping cough, pneumonia/pneumococcal diseases, meningococcal disease, hepatitis B and human papillomavirus. Notably, some of these vaccines have previously been shown to transiently induce immune activation and/or affect the HIV reservoir. For instance, a study involving the administration of the influenza vaccine in PWH on ART with suppressed viral load showed HIV RNA transcription can occur in the week following vaccination9. The authors also noted enhanced immune activation (as defined by CD38 and HLA-DR expression) during the four weeks after vaccination. Similarly, another study investigating the effect of the pneumococcal vaccine on ART-treated PWH with suppressed viral loads observed a transient increase in plasma HIV RNA levels post-vaccination which returned to undetectable levels within four weeks25. Moreover, previous work from some of the co-investigators of this current grant application also demonstrated that the influenza vaccine can disproportionately increase HIV proviral burden in influenza-specific CD4+ T cells of ART-treated PWH with suppressed viral loads, suggesting the ability of vaccination to affect the HIV reservoir26.

A significant gap in our knowledge is whether COVID-19 vaccines, especially with its novel mRNA-based platform, may have any impact on ongoing chronic inflammation and other immune dysregulation that can exacerbate co-morbidity incidence or affect the dynamics of the HIV reservoir in PWH.

A significant gap in our knowledge is whether COVID-19 vaccines can induce protective and robust immune responses both in the short-term and long-term, particularly in specific subgroups with well-described, diminished immunocompetence. This is a critical issue to address as agencies including NACI have expressed concerns around efficacy in the context of immunodeficiency. Current NACI recommendation states that "currently, there are no data on COVID-19 vaccination in individuals who are immunosuppressed" and that since "[t]he relative degree of immunodeficiency in individuals who are immunocompromised is variable depending on the underlying condition, the progression of disease and use of medications that suppress immune function... the balance of benefits and risks must be made on a case-by-case basis". Moreover, there is suggestion that immunosenescence and older age may have important implications as evidenced by a reduced efficacy with a wide confidence interval with both vaccines in participants older than 65. Another significant gap in our knowledge is that the investigators do not know whether COVID-19 vaccines may have any impact on ongoing chronic inflammation and other immune dysregulation that can exacerbate co-morbidity incidence or affect the dynamics of the HIV reservoir. Importantly, neither of these knowledge gaps are likely going to be evaluated by vaccine sponsors.

STUDY OBJECTIVES To evaluate the effect of COVID-19 vaccines on generating SARS-CoV-2 specific immune response, inducing systemic immune activation and affecting HIV viral reservoirs in PWH.

Hypotheses:

Primary: PWH will exhibit diminished immune response towards COVID-19 vaccines in terms of robustness and durability of immune response.

Secondary: COVID-19 vaccines will adversely affect immune activation and HIV reservoirs in PWH.

STATISTICAL ANALYSIS Baseline characteristics will be examined to assess the comparability of the participants in the study arms. Continuous variables such as age and CD4+ T cell count will be described in terms of medians and interquartile ranges. Categorical variables such as gender and race will be described with proportions.

Analyses between HIV-positive and HIV-negative groups will be using 2- sample Student's t-test or Wilcoxon test if there is a deviation of normality. Two-sided 95% confidence intervals will be obtained by performing logarithmic transformations of titers calculating the 95% confidence interval with reference to Student's t-distribution, and then exponentiating the limits of the confidence intervals. Attempts will be made to look for trends between HIV subgroups listed above.

* medication within the past 6 months (topical steroids are allowed)
* For HIV-negative participants: immune-compromising conditions or on medication which suppresses the immune response

STUDY DESIGN This is a prospective, non-randomized observational study to examine SARS-CoV-2 vaccine immunogenicity, immune activation and HIV reservoirs in people with HIV infection in comparison with HIV-negative individuals, in those aged 55 or more.

As Canada is currently rolling out COVID-19 vaccines, the two most imminent vaccines are mRNA vaccines. These are the Pfizer-BioNTech COVID-19 vaccine given 3 weeks apart and the Moderna COVID-19 vaccine given 4 weeks apart. Given the unique storage requirements of these vaccines, it is expected that the Moderna vaccine will be used primarily in primary care clinics such as Maple Leaf Medical Clinic, Toronto. However, the protocol will also allow observational study of individuals being administered with the Pfizer-BioNTech vaccine if it is also available. The investigators predict general availability of both vaccines to the primary care population by March 1, 2021. Vaccination will occur as per clinical and public health guidelines. COVID-19 vaccines will not be administered as a part of this research study.

Study duration: This is a single site longitudinal study where 75 participants in total are followed over 48 weeks with blood draws and saliva sampling. Evaluations will be taken at screening, baseline and at 8 additional time points during the study. Details on screening and follow-up visits are outlined in section 4.4 Sampling.

Recruitment plan

A total of 75 participants will be recruited for the study. The clinical research coordinator will perform chart review with the Principal Investigator's oversight to contact potential study participants who meet the eligibility criteria. The breakdown of study arms is described here:

• PWH Immune responders (n= 35): undetectable viral load for 1+ year, CD4 >500/uL, CD4/CD8 ratio >1 including individuals with a historical, low CD4 nadir

• PWH Immune non-responders (n= 10): undetectable viral load, CD4 <350/uL or CD4/CD8 ratio <0.75 for 1+ year

• PWH Low-level viremics (n= 10): low-level viremia (<1,000 copies/mL) for 1+ year, any CD4, any CD4/CD8 ratio

• HIV-negative control (n= 20): age and sex matched

As enrolment progresses, the investigators will attempt to increase numbers in the PWH Immune non-responders and PWH Low-level viremics arms, as appropriate and feasible.

Screening Participants will be assessed to gauge interest in participating in the clinical trial and appropriateness for the study based on inclusion and exclusion criteria. Database search will also focus on optimizing demographic diversity based on race/ethnicity and sex/gender. Participants who are interested in the study and who satisfy the inclusion and exclusion criteria will be given the consent form to review and any questions will be answered. The screening visit will take place within 90 days prior to the baseline visit.

Routine blood work will be performed at the screening visit including hematology, biochemistry, sexually transmitted infections and C-reactive protein. In addition to the routine blood work, the following will be performed in HIV-positive participants: CD4 count, viral load, CD4/CD8 ratio. In addition to the routine blood work, the following will be performed in HIV-negative participants: HIV test.

Sampling:

Visit Time Date Research Specimens

1. Screening* Up to 90 days before baseline
2. Baseline Up to 24 hours before vaccine 13 blood tubes (113.5mL), saliva

1st dose of COVID-19 vaccine (clinical procedure; not a part of this research study) 3 Follow-up 1 10 days after 1st vaccine 7 blood tubes (62.5mL) 4 Follow-up 2 21 days after 1st vaccine 7 blood tubes (62.5mL) 5 Follow-up 3 28 days after 1st vaccine 13 blood tubes (113.5mL), saliva 2nd dose of COVID-19 vaccine (clinical procedure; not a part of this research study) 6 Follow-up 4 7 days after 2nd vaccine 7 blood tubes (62.5mL), saliva 7 Follow-up 5 14 days after 2nd vaccine 7 blood tubes (62.5mL) 8 Follow-up 6 28 days after 2nd vaccine 7 blood tubes (62.5mL) 9 Follow-up 7 24 weeks after 1st vaccine 13 blood tubes (113.5mL), saliva 10 Follow-up 8* 48 weeks after 1st vaccine 13 blood tubes (113.5mL)

The figure above describes all study visits and specimens collected at each visit. Participants must provide copy of vaccination card confirming they received the COVID-19 vaccine. Baseline visit (V1) is defined as specimen collection up to 24 hours prior to receiving the first dose of the COVID-19 vaccine. All other subsequent visits will take place +/- 3 days of the indicated days. It should be noted that V3 (21 days post-prime vaccine visit) must take place prior to receiving the 2nd dose of the vaccine, regardless of whether the participants receive Moderna or Pfizer-BioNTech vaccine.

In the event that a participant does not get their booster at the scheduled date, all post booster time points will be adjusted according to the time of the booster dose. For example, if a participant came to get their Moderna booster at 35 days post-prime instead of the scheduled time of 28 days post-prime for reasons beyond their control, then V4 and V5 time points would be adjusted accordingly. The investigators will allow a delay for the booster in this study in order for a participant to remain in the study protocol, as it is expected that immunity should still be obtained with a booster at a delayed time point. Moreover, if the second dose is delayed by more than 2 weeks (i.e. Ontario's current push for delaying the second dose by up to 16 weeks), the investigators will add in one visit before the scheduled second dose (up to 7 days before second dose). Study visits will therefore be revised for people with > 2 weeks of delayed second dose as the following:

Visit Time Date Research Specimens

1. Screening* Up to 90 days before baseline
2. Baseline Up to 24 hours before vaccine 13 blood tubes (113.5mL), saliva

1st dose of COVID-19 vaccine (clinical procedure; not a part of this research study) 3 Follow-up 1 10 days after 1st vaccine 7 blood tubes (62.5mL) 4 Follow-up 2 21 days after 1st vaccine 7 blood tubes (62.5mL) 5 Follow-up 3 28 days after 1st vaccine 7 blood tubes (62.5mL), saliva 6 Follow-up 4 7 days before delayed 2nd vaccine 13 blood tubes (113.5mL), saliva 2nd dose of COVID-19 vaccine (clinical procedure; not a part of this research study) 7 Follow-up 5 7 days after 2nd vaccine 7 blood tubes (62.5mL), saliva 8 Follow-up 6 14 days after 2nd vaccine 7 blood tubes (62.5mL) 9 Follow-up 7 28 days after 2nd vaccine 7 blood tubes (62.5mL) 10 Follow-up 8 24 weeks after 1st vaccine 13 blood tubes (113.5mL), saliva 11 Follow-up 9* 48 weeks after 1st vaccine 13 blood tubes (113.5mL)

Given the frequent number of blood draws, participants will still be invited to remain in the study if they miss visits.

It is possible that some participants may be offered a third booster dose of vaccine according to new recommendations made by Ontario and Canadian vaccine agencies due to potential vaccine waning by 6 months or other underlying immunosuppression (e.g., chemotherapy). If a participant does receive a booster dose, they will be invited to provide a blood draw (7 blood tubes) and saliva within 7 days of the 3rd booster and then 1 and 3 months afterward. If these visits are close in time to the same time points of the already scheduled follow up visits in the above chart by one week, then the investigators will use that blood draw also as the follow up visits.

Assignment of Participant Identification Numbers Each participant who consents will be assigned a unique participant identification number (PID), which identifies the participant for all study-related procedures. PIDs are a combination of four-digit site number plus 3-digit participant number starting with 001 (e.g., 3001-001). Once assigned, PIDs cannot be reused for any reason.

Clinical evaluations:

Screening visit: Participants will be assessed to gauge interest in participating in the study and appropriateness for the study based on inclusion and exclusion criteria. Participants who are interested in the study and who satisfy the inclusion and exclusion criteria will be given the consent form to review and any questions will be answered. Clinical evaluations will include a medical history (to be conducted by the research coordinator through chart review with the Principal Investigator's oversight) and routine blood work in addition to viral load, CD4 count, CD4/CD8 ratio for HIV-positive participants and HIV test for HIV-negative participants. Concomitant medication history and cART regimen will be documented at each visit. Documentation of COVID-19 infection will also be assessed: This is documented as occurring in participants who had at least two of the following symptoms: fever (temperature ≥38C), chills, myalgia, headache, sore throat, or new olfactory or taste disorder, or as occurring in those who had at least one respiratory sign or symptom (including cough, shortness of breath, or clinical or radiographic evidence of pneumonia) and at least one nasopharyngeal swab, nasal swab, or saliva sample (or respiratory sample, if the participant was hospitalized) that was positive for SARS-CoV-2 by reverse-transcriptase-polymerase-chain-reaction (RT-PCR) test. Demographics: Demographic information (date of birth, gender, race) will be recorded at Screening.

Vaccination: Participants will be administered COVID-19 vaccines according to standard specifications provided by the vaccine manufacturers. Vaccination is not a research study visit, but rather administered as per clinical and public health guidelines. The vaccine most likely to be administered due to availability and storage requirements will be the Moderna COVID-19 vaccine, which will be administered on day 0 and week 4 (28 days later). It is also possible that the Pfizer-BioNTech COVID-19 vaccine will be available which will be administered by the primary care provider on day 0 and week 3 (21 days later). The date of vaccination and vaccine product (Moderna or Pfizer-BioNTech) will be documented.

COLLECTION OF SPECIMENS:

As this is an observational study, only specimens and clinical information will be collected.

Baseline (V2):

Up to 24 hours prior to receiving the vaccination, the following will be obtained: Confirmation of cART regimen; A saliva specimen using a salivette tube to be given to participant and returned to clinical study coordinator after one minute; Venipuncture of 1 SST tube, 2 EDTA, and 10 ACD tubes (113.5 ml blood)

Day 10 Post-prime (V3):

Assessment of new or continuing concomitant medications, including cART regimen; Assessment if developed COVID-19 infection; Venipuncture of 1 SST, 2 EDTA and 4 ACD tubes (62.5 ml blood); Inquire about immediate vaccine reactogenicity

Day 21 Post-prime (V4):

Assessment of new or continuing concomitant medications, including cART regimen; Assessment if developed COVID-19 infection; Venipuncture of 1 SST, 2 EDTA and 4 ACD tubes (62.5 ml blood)

Day 28 Post-prime (V5):

Assessment of new or continuing concomitant medications, including cART regimen; A saliva specimen using a salivette tube to be given to participant and returned to clinical study coordinator after one minute; Venipuncture of 1 SST tube, 2 EDTA, and 10 ACD tubes (113.5 ml blood)

Day 7 Post-booster (V6 or V7 if delayed second dose):

Assessment of new or continuing concomitant medications, including cART regimen; Assessment if developed COVID-19 infection; Saliva specimen; Venipuncture of 1 SST, 2 EDTA and 4 ACD tubes (62.5 ml blood); Inquire about immediate vaccine reactogenicity

Day 14 Post-booster (V7 or V8 if delayed second dose ):

Assessment of new or continuing concomitant medications, including cART regimen; Assessment if developed COVID-19 infection; Venipuncture of 1 SST, 2 EDTA and 4 ACD tubes (62.5 ml blood)

Day 28 Post-booster (V8 or V9 if delayed second dose ):

Assessment of new or continuing concomitant medications, including cART regimen; Assessment if developed COVID-19 infection; Venipuncture of 1 SST, 2 EDTA and 4 ACD tubes (62.5 ml blood)

Week 24 Post-prime (V9 or V10 if delayed second dose ):

Assessment of new or continuing concomitant medications, including cART regimen; Assessment if developed COVID-19 infection; Saliva specimen; Venipuncture of 1 SST tube, 2 EDTA, and 10 ACD tubes (113.5 ml blood)

Week 48 Post-prime (V10 or V11 if delayed second dose ):

Assessment of new or continuing concomitant medications, including cART regimen; Assessment if developed COVID-19 infection; Venipuncture of 1 SST tube, 2 EDTA, and 10 ACD tubes (113.5 ml blood)

If the second dose is delayed by more than 2 weeks, an additional study visit will be scheduled immediately (up to 3 days) before the second dose. This visit will be visit #6 where a total of 1 SST tube, 2 EDTA, and 10 ACD tubes (113.5ml blood) will be collected in addition to saliva specimen. All subsequent visits will be adjusted accordingly whereby the original V6 becomes V7, V7->V8 and so forth, ending with V10->V11.

Research projects:

Saliva and a subset of blood specimens will go to the University of Toronto. Specimens going to the University of Toronto and affiliated hospitals will be centrally processed in the Ostrowski lab at the Medical Sciences building, University of Toronto and stored in the Ostrowski lab. Specimens for the NIH will be directly shipped from Maple Leaf Medical Clinic to the Chun lab at NIH, Bethesda, MD, USA. Saliva assays will be done by the Gommerman lab at the University of Toronto. Serological assays will be done by the Gingras lab at Mount Sinai Hospital, which is affiliated with the University of Toronto. Neutralization assays and T cell immune responses to COVID-19 will be performed at the Ostrowski lab. The IPDA assay will be done at the Ostrowski lab in collaboration with Brad Jones (Cornell University). Samples sent to the NIH will be stored in the Chun lab and the Chun lab will perform viral reservoir assays, and immune activation assays. The Moir lab will perform B cell immune studies. All laboratories have extensive experience in managing human specimens from processing to storage. All samples leaving the Maple Leaf Clinic are de-identified.

The following assays will be performed in the following labs:

Dr. Mario Ostrowski's group:

The Ostrowski lab has developed expertise in developing an in-house, micro-neutralization assay of live SARS-CoV-2 virus. In addition, his lab has provided pre-clinical studies on the development of a Canadian COVID-19 mRNA vaccine in collaboration with Providence Therapeutics in Canada27. The lab routinely is performing SARS-CoV-2 neutralization assays for a number of investigators. The lab also has characterized T cell immune responses in COVID-19 infection and will use T cell ELISPOT assays to determine T cell immune responses to the vaccine antigens28. The lab is mainly an HIV lab, and in collaboration with Dr. R. Brad Jones at Cornell University, will perform the intact proviral DNA assays. The Jones lab has extensive experience in designing an in-house assay which he will share the protocol at U of Toronto, to expedite data analysis. They have both published on this assay29. The following assays will be performed at W0, W24, W48: Neutralization titer to SARS-CoV-2 (plaque reduction microneutralization assay); T cell ELISPOT to SARS-CoV-2 IPDA (intact proviral DNA assay).

Dr. Tae-Wook Chun's group:

Dr. Chun's program focuses on 1) delineating the role of viral reservoirs in the pathogenesis of HIV disease; 2) examining host and viral factors that contribute to the maintenance of HIV reservoirs; and 3) developing therapeutic strategies aimed at achieving durable virologic control in infected individuals in the absence of antiretroviral therapy. Dr. Chun's laboratory will conduct multiple HIV viral reservoir assays, extensive immune phenotyping of T cells, and profiling of soluble biomarkers.

Dr. Susan Moir's group:

The primary focus of Dr. Moir's research program is to study the role of B cells in the pathogenesis of HIV disease, with the ultimate goal of filling gaps in knowledge regarding humoral immunity against the virus. This knowledge is critical to the development of an effective antibody-based vaccine and for advancement of immunotherapeutic interventions in HIV-infected individuals. Dr. Moir will primarily focus on longitudinal B-cell/plasmablast phenotyping and antigen-specific responses and B-cell/memory phenotyping and antigen-specific responses.

Dr. Jennifer Gommerman's group:

Dr. Gommerman leads a COVID-19 team that is looking into salivary mucosal responses to SARS-CoV-2, and in particular the IgA response, which is felt to be crucial to protect from infection and carriage of the virus. Her team will use collected saliva samples to test for IgA response to SARS-CoV-2 S and RBD. Her lab has developed sensitive and specific assays in house to determine mucosal immunity to the SARS-CoV-2 virus30. It is unknown whether the current COVID-19 vaccines induce any immunity at the mucosal level. The following assays will be done at W0, 5, 24: Salivary IgA to SARS-CoV-2 S, RBD and NP.

Dr. Anne-Claude Gingras' group:

Dr. Anne-Claude Gingras is an expert in protein interaction and high throughput studies and her group has developed SARS-CoV-2 spike and Receptor Binding Domain (RBD) and nucleocapsid protein ELISA tests (IgG, IgA, IgM) on a robotic platform that can be scaled up to test thousands of samples per day. She has also developed an ELISA-based surrogate assay that can predict neutralization ability of serum to SARS-CoV-2 and optimized a lentivirus-based spike neutralization assay30,31. The following assays will be done at all time points and screening: Serum IgG to SARS-CoV-2, nucleocapsid, and RBD domain. The presence of these antibodies at baseline will indicate prior SARS-CoV-2 and will be an exclusion criterion. The COVID vaccines only induce antibodies to SARS-CoV-2 spike protein and responders should develop antibodies to spike and RBD, but not to the nucleocapsid. Antibodies to the nucleocapsid would indicate immune response to infection rather than to the vaccine.

REB review and approval- conduct of the study The site will obtain approval for the study protocol and, consent form prior to the start of the study from the University of Toronto Research Ethics Board REB. The REB will review all appropriate study documentation to safeguard the rights, safety, and well-being of the participants. The study will be conducted only after ethics approval has been obtained. A copy of the protocol (including protocol amendments), all versions of informed consent forms, other information to be completed by participants such as survey instruments or questionnaires, and any proposed advertising/ recruitment materials must be reviewed and approved by the REB of each participating center prior to implementation of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants will fall into any of the HIV-positive arms or the HIV-negative control arm. Inclusion criteria for HIV-positive participants are:

  * Ability to provide signed written informed consent
  * Documented HIV diagnosis for 1+ year
  * Antiretroviral therapy for 1+ year
  * 55 years of age or older
  * Good general health as shown by medical history and screening laboratory tests at the screening visit:

    * Hemoglobin ≥ 85 g/L White blood cell (WBC) count = 3300 to 12,000 cells/mm3
    * Total lymphocyte count ≥ 800 cells/mm3
    * Platelets = 50,000 to 550,000/mm3
    * Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase < 5 times the institutional upper limit of normal (ULN); creatinine (Cr) ≤ institutional upper limit of normal; creatine phosphokinase (CPK) ≤ 2 times the institutional upper limit of normal not related to physical exertion

Inclusion criteria for HIV-negative participants are:

* Ability to provide signed written informed consent
* Negative HIV test at the screening visit
* 55 years of age or older
* Stable clinical status and absence of acute illnesses as shown by medical history and screening laboratory tests at the screening visit:

  * Hemoglobin ≥ 85 g/L White blood cell (WBC) count = 3300 to 12,000 cells/mm3
  * Total lymphocyte count ≥ 800 cells/mm3
  * Platelets = 50,000 to 550,000/mm3
  * Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase < 5 times the institutional upper limit of normal (ULN); creatinine (Cr) ≤ institutional upper limit of normal; creatine phosphokinase (CPK) ≤ 2 times the institutional upper limit of normal not related to physical exertion

Exclusion Criteria:

* There will be no exclusion criteria based on gender/gender identity, ethnoracial composition, language, socioeconomic status, mode of HIV acquisition or sexual orientation/identity. Any participant who requires language interpretation can and will be accommodated for by the participation of translators, either at the patient's choice and/or with the assistance of the translator services provided by local ASO organizations. Exclusion criteria include the following:

  * Participants who would have difficulty participating in a trial due to non-compliance
  * Participants with a history of anaphylaxis reaction to the COVID-19 vaccine components
  * Participants with any of the following abnormal laboratory results at the screening visit:

    * Hemoglobin < 85 g/L
    * Lymphocyte count < .750 X109/L
    * Platelet count < 50 X109/L or > 550 X109/L
    * AST or ALT > 5X the upper limit of normal
    * Creatinine > 250 µmol/L
  * Participant with a malignancy or undergoing chemotherapy
  * Participant with other significant underlying disease (non-HIV-1) that might impinge upon disease progression or death
  * Active infection with hepatitis virus (HAV, HBV, HCV) or tuberculosis
  * Prior surgery or radiation therapy within 30 days of study screening or receipt of any other experimental compound within 30 days of signing informed consent
  * Any concurrent condition requiring the continued use of immunoglobulin, antineoplastic agents, glucocorticoids (other than corticosteroid nasal spray for allergic rhinitis; topical or ophthalmic corticosteroids for acute, uncomplicated dermatitis or conjunctivitis; over the counter medications for acute, uncomplicated dermatitis for treatment period not longer than 14 days) or other immunomodulator medications (other than NSAIDS which will be allowed for any length of time)
  * Receipt of any blood product within 3 months prior to screening
  * Receipt of any vaccine within 1 month prior to screening
  * Active drug or alcohol use/dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
  * Any illness or conditions including acute illnesses that, in the opinion of the investigator, may affect the safety of the participant or the evaluation of any study endpoints
  * Any other conditions judged by the investigator that would limit the evaluation of a participant
  * Positivity for sexually transmitted infections at the screening visit
  * Use of any unproven registered and unregistered treatments for COVID-19; Administration of immunoglobulins and/ or any blood products within the three months preceding the planned administration of the vaccine candidate
  * Any confirmed or suspected immunosuppressive or immunodeficient state (except HIV infection for Group-3), asplenia, recurrent severe infections and chronic use (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
  * For HIV-negative participants: immune-compromising conditions or on medication which suppresses the immune response.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People diagnosed with HIV (1+ year), 55 years of age or older, on antiretroviral therapy for 1+ year with good general health as per medical history and lab tests. HIV negative individuals, 55 years old or older with stable clinical status, without acute illnesses as per medical history and lab tests will also be recruited for control.
  Blood and saliva sampling at described timepoint prior to 1st dose of COVID-19 vaccination and after the second dose of the COVID-19 vaccination. Evaluations will be taken at screening, baseline and at 8 additional time points during the study. 75 participants will be followed over 48 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Primary | Week 24
  Serum SARS-CoV-2 Neutralization assay (plaque reduction microneutralization assay) will be compared between HIV-positive and negative groups.

SECONDARY OUTCOMES:
Neutralization titers | Baseline and Week 48
  Neutralization titers in serum against live SARS-CoV-2
IgG; RBD; NCP | Weeks 0, 1, 2, 5, 6, 8, 24 and 48
  IgG levels to spike (S) protein, receptor binding domain (RBD) and nucleocapsid protein (NP)
T cell | Week 24 and Week 48
  T cell responses against the S protein at baseline
Salivary IgA | Week 5 and Week 24
  Salivary IgA levels to S protein and RBD
COVID-19 Infection | Up to week 48
  Rates of COVID-19 infection
Provirus | baseline, Week 24 and Week 48
  Integrated (IPDA) and non-integrated provirus
Activation Parameters | Weeks 0, 1, 2, 5, 6, 8, 24 and 48
  Activation parameters of T cells and B cells via flow cytometry
Cytokine and Chemokine | Weeks 0, 1, 2, 5, 6, 8, 24 and 48
  Inflammatory cytokine and chemokine levels via multiple PCR assays
B-cell/plasmablast | Weeks 0, 1, 2, 5, 6, 8, 24 and 48
  B-cell/plasmablast phenotyping and antigen-specific responses
B-cell/memory | Weeks 0, 1, 2, 5, 6, 8, 24 and 48
  B-cell/memory phenotyping and antigen-specific responses

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ostrowski, MD, Principal Investigator — University of Toronto
Locations (1):
- Maple Leaf Medical Clinic, Toronto, Ontario, Canada